CLINICAL TRIAL: NCT00353392
Title: Q-Switched Nd:YAG in Macular Amyloidosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: src-ost-1359
Record Dates: First submitted 2006-07-17; First posted 2006-07-18 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2006-11

CONDITIONS: Macular Amyloidosis
MeSH Terms: interventions — Laser Therapy

INTERVENTIONS:
Device: Laser Therapy

SUMMARY:
The purpose of this study is to determine whether Q-Switched Nd:YAG Laser therapy are effective in reduction of Cutaneous macular amyloidosis.

DETAILED DESCRIPTION:
We treat the macular amyloidosis cases by Q-Switched Nd:YAG Laser and compare the before and after treatment situation by the photos and colorimetric assessment.

ELIGIBILITY:
Inclusion Criteria:

* Macular amyloidosis confirmed cases

Exclusion Criteria:

* Pregnancy and breast feeding
* Over 18 years old

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2006-03; Primary Completion 2006-07 (Actual); Study Completion 2006-08

PRIMARY OUTCOMES:
Visual and colorimetric assessment

CONTACTS AND LOCATIONS:
Overall Officials: Nima Ostovari, M.D., Study Director — Shahid Beheshti University of Medical Sciences; Parviz Toossi, MD, Study Chair — Shaheed Beheshti Medica University
Locations (1):
- Skin Research Center, Shaheed Beheshti Medical University, Tehran, Iran